CLINICAL TRIAL: NCT01272869
Title: Clinical Investigation of Filter Improvement for New Filter to Ostomy Bags
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP211OC
Record Dates: First submitted 2010-12-14; First posted 2011-01-10 (Estimated); Results first posted 2012-12-31 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-11

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sensura (Active Comparator): SenSura is the reference product and the product is already commercially available
  Interventions: Device: SenSura
- Morfeus (Experimental): The test product is the product with the proposed new filter (Morfeus)
  Interventions: Device: Morfeus

INTERVENTIONS:
Device: SenSura — The ostomy bag filter will be tested for a period of 14 days
  Arms: Sensura
Device: Morfeus — The new ostomy bag filter will be tested for a period of 14 days
  Arms: Morfeus

SUMMARY:
The aim of the current clinical investigation is to evaluate a new filter

DETAILED DESCRIPTION:
The filter has been developed in order to significantly reduce problems with ballooning and other problems related to filter performance in people with a stoma.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age and have full legal capacity.
* Have given written informed consent.
* Be able to fill in the Case Report Form.
* Be ileostomy operated and have had a stoma for at least 6 months.
* Experience ballooning at least once per week.
* Be able to manage the bags themselves (application, removal).
* Be able to use a flat base plate.
* Have a stoma with a diameter less than 60 mm

Exclusion Criteria:

* Persons who irrigate
* Currently suffer from peristomal skin problems (i.e. bleeding or broken skin).
* Currently receiving or have within the past 2 months received radio- and/or chemotherapy.
* Pregnant or breastfeeding.
* Participate in other test at the same time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Carter, MSc, Study Chair — Coloplast A/S
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were recruited from a user data base in Denmark.
Pre-assignment Details: 20 subjects were enrolled and randomized in the study.
Groups:
- Sensura First; Then Morfeus: The reference product is the SenSura product which is already commercially available
- Morfeus First; Then Sensura: The test product with the Morfeus filter is the test product with the proposed new filter.
Period: Period 1 (14 Days)
Arm/Group | Sensura First; Then Morfeus | Morfeus First; Then Sensura
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Period 2 (14 Days)
Arm/Group | Sensura First; Then Morfeus | Morfeus First; Then Sensura
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sensura: The reference product is the SenSura product which is already commercially available
- Total: Total of all reporting groups
Arm/Group | Sensura | Morfeus | Total
Number analyzed (Participants) | 10 | 10 | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 59 (13) | 61 (10) | 60 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 4 | 9 | 13

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Ballooning in the Morfeus and the Sensura Filter Test Period.
Description: Data will not be recorded at specific time points due to individual changing patterns (1-2 bags per day). Study subjects will fill out the Case Report Form (CRF) by themselves when changing bag. The subject is asked in the CRF among others the reason for changing bag (e.g. ballooning). Subjects will change bag according to their normal routine or when deemed appropriate. They are advised to change bag if it is filled with air and the air cannot be released through the filter within a specified time period.
Time Frame: Daily or at every change of bag in a period of a maximum of 28 days
Population: Intention to treat (ITT)
Measure: Number; unit: percentage bags with ballooning
Units Other Than Participants: Bags
Arm/Group | Sensura | Morfeus
Number analyzed (Participants) | 20 | 20
Number analyzed (Bags) | 156 | 146
percentage bags with ballooning | 55 | 26

ADVERSE EVENTS:
Arm/Group | Sensura | Morfeus
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 3/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensura (N=20) | Morfeus (N=20)
Abscess in the buttock (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensura (N=20) | Morfeus (N=20)
Pristomal skin redness (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Sleep disruption (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes